CLINICAL TRIAL: NCT02701855
Title: Retina Microvascular Remodeling and Cognitive Function In Hypertension : Eyebrain
Brief Title: Retina Microvascular Remodeling and Cognitive Function In Hypertension
Acronym: EYEBRAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cardiometabolism and Nutrition, France (Other)
Collaborators: Fondation de Recherche sur l'Hypertension Artérielle (Other)
Responsible Party: Sponsor
Other Study IDs: 14DRM_EYEBRAIN
Record Dates: First submitted 2015-08-04; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension; Mild Cognitive Impairment
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction | interventions — Neuropsychological Tests; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hypertension and progressive MCI: 50 subjects will perform brain and aorta RMI, blood test, cognitive tests and adaptative optics.
  Interventions: Behavioral: Cognitive tests; Biological: Blood test; Radiation: Brain and aorta RMI; Other: Adaptative optics
- Hypertension and stable MCI: 50 subjects will perform brain and aorta RMI, blood test, cognitive tests and adaptative optics.
  Interventions: Behavioral: Cognitive tests; Biological: Blood test; Radiation: Brain and aorta RMI; Other: Adaptative optics
- Hypertension, without MCI: 60 subjects will perform brain and aorta RMI, blood test, cognitive tests and adaptative optics.
  Interventions: Behavioral: Cognitive tests; Biological: Blood test; Radiation: Brain and aorta RMI; Other: Adaptative optics

INTERVENTIONS:
Behavioral: Cognitive tests — Cognitive tests include:
  * The MMSE (Mini Mental State Examination)
  * Free and Cued Selective Recall Reminding Test (FCSRT).
  * Executive functions (fluencies, TMT A and B, span).
  * Tests of verbal fluency (literal and category)
  * Digit symbol substitution test or Wechsler adult intelligence scale (W.A.I.S)
  * The Clinical Dementia Rating Scale
  * The IADL scale evaluates autonomy.
  * Geriatric Depression screening Scale (GDS)
Biological: Blood test — A blood test will be performed in order to collect following parameters: Urea, BUN, Creatinine, Potassium, Sodium, hematocrit, hsCRP, NFS, Pq, LDL-C, HDL-C, Triglycerides, Lp(a), Lp-PLA2 as well as fasting glucose, HbA1C and microalbuminuria
Radiation: Brain and aorta RMI — A magnetic resonance imaging exam will be performed at the Neuroimaging Research Center of the Pitié-Salpêtrière Hospital. This exam will be optimized to fit in 30 minutes. Indeed brain 3D T1 and T2 FLAIR imaging lasts 15 minutes while cine and velocity encoded imaging of the aorta lasts 15 minutes.
Other: Adaptative optics — The retina adaptative optic imaging will be performed at the "Unité de prevention des maladies cardiovasculaires" Pitié Salpetrière Hospital. This exam lasts 10 minutes including patient positioning and imaging.

SUMMARY:
This study aims to determine the relationships between retina micro-vascular remodeling and cognitive function in hypertensive patients.

The study plans to enrol 160 patients (100 patients with mild cognitive impairment -MCI- and 60 without MCI).

DETAILED DESCRIPTION:
Our project stands on physiopathological and cognitive angles, and is mainly based on the major role of large and small arteries elasticity on cognitive aging. It will benefit from the recent innovative accurate and non invasive techniques such as MRI for central large arteries and adaptative optics for retina arterioles imaging.

Study population is the following:

* 60 patients with hypertension and no MCI,
* 50 patients with hypertension and stable MCI, without dementia
* 50 patients with hypertension and progressive MCI, without dementia

Every patients will perform a medical interview and examination, an MRI (brain + aorta), adaptative optics imaging, a cognitive tests and a blood test.

Primary outcome is to determine the relationships between retina micro-vascular remodeling and cognitive function in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or more
2. hypertension (BP ≥140/90 mmHg and/or antihypertensive treatment)
3. Signed informed consent by the patient
4. Sufficient mastery of the French language to perform neuropsychological tests

Exclusion Criteria:

1. Impossibility to visualize the retinal : severe cataract
2. Dementia (defined by MMSE<20)
3. Clinical stroke
4. Severe or resistant Hypertension
5. Hypertension treated with more than 3 different pharmacological classes
6. any other disease that may interfere with the assessment of cognitive disorders (epilepsy, Parkinson's disease, major depression, schizophrenia, manic-depressive)
7. Enrolment in a therapeutic trial that could interfere with the main objective
8. Less than 4 years of formal education
9. Illiterate, unable to read, write or count
10. major physical problems that may interfere with the tests (sight, hearing, ...)
11. Short term life threatening disease
12. Non-affiliation to a healthcare system
13. Consent refusal
14. Contraindication to MRI including claustrophobia, metallic devices, pacemaker, mechanical valve implanted before 1985, and nursing, as well as technical contra-indication: patient diameter > 70 cm or/and weight > 250 kg

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients' recruitment will be carried out in two centers to ensure inclusion of both patients: 1) with hypertension and without cognitive impairment, 2) with hypertension and with mild cognitive impairment (without dementia) including patients with stable MCI and converters.
  Population size: 160 patients:
  * 60 patients with hypertension and no MCI,
  * 50 patients with hypertension and stable MCI, without dementia
  * 50 patients with hypertension and progressive MCI, without dementia
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Relationships between retina micro-vascular remodeling and cognitive function in hypertensive patients. | September 2017

SECONDARY OUTCOMES:
• Associations between cognitive function and proximal aortic stiffness indices estimated from MRI images. | September 2017
• Associations between retina arteriolar remodelling and cerebrovascular lesions (infarcts, lacuna, and white matter lesions) quantified from MRI images. | September 2017
• Associations between retina arteriolar remodelling and neurodegenerative lesions (hippocampus atrophy) quantified from MRI images. | September 2017
• Associations between proximal aortic stiffness and cerebrovascular lesions (infarcts, lacuna, and white matter lesions) quantified from MRI images. | September 2017
• Associations between proximal aortic stiffness and neurodegenerative lesions (hippocampus atrophy) quantified from MRI images. | September 2017
• Associations between retina arteriolar remodelling and proximal aortic stiffness indices. | September 2017

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de prévention des maladies cardiovasculaires Pôle Cardiologie/Métabolisme Hôpital Pitié-Salpétriêre, APHP, 83 bd de l'hôpital,, Paris, France

REFERENCES:
- [Background] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- [Background] Luchsinger JA, Reitz C, Honig LS, Tang MX, Shea S, Mayeux R. Aggregation of vascular risk factors and risk of incident Alzheimer disease. Neurology. 2005 Aug 23;65(4):545-51. doi: 10.1212/01.wnl.0000172914.08967.dc. PMID 16116114
- [Background] Launer LJ, Ross GW, Petrovitch H, Masaki K, Foley D, White LR, Havlik RJ. Midlife blood pressure and dementia: the Honolulu-Asia aging study. Neurobiol Aging. 2000 Jan-Feb;21(1):49-55. doi: 10.1016/s0197-4580(00)00096-8. PMID 10794848
- [Background] Qiu C, Winblad B, Fratiglioni L. The age-dependent relation of blood pressure to cognitive function and dementia. Lancet Neurol. 2005 Aug;4(8):487-99. doi: 10.1016/S1474-4422(05)70141-1. PMID 16033691
- [Background] Perlmutter LS, Barron E, Saperia D, Chui HC. Association between vascular basement membrane components and the lesions of Alzheimer's disease. J Neurosci Res. 1991 Dec;30(4):673-81. doi: 10.1002/jnr.490300411. PMID 1787541
- [Background] Hardy JA, Mann DM, Wester P, Winblad B. An integrative hypothesis concerning the pathogenesis and progression of Alzheimer's disease. Neurobiol Aging. 1986 Nov-Dec;7(6):489-502. doi: 10.1016/0197-4580(86)90086-2. PMID 2882432
- [Background] Vagnucci AH Jr, Li WW. Alzheimer's disease and angiogenesis. Lancet. 2003 Feb 15;361(9357):605-8. doi: 10.1016/S0140-6736(03)12521-4. PMID 12598159
- [Background] Hanon O, Haulon S, Lenoir H, Seux ML, Rigaud AS, Safar M, Girerd X, Forette F. Relationship between arterial stiffness and cognitive function in elderly subjects with complaints of memory loss. Stroke. 2005 Oct;36(10):2193-7. doi: 10.1161/01.STR.0000181771.82518.1c. Epub 2005 Sep 8. PMID 16151027
- [Background] Redheuil A, Yu WC, Wu CO, Mousseaux E, de Cesare A, Yan R, Kachenoura N, Bluemke D, Lima JA. Reduced ascending aortic strain and distensibility: earliest manifestations of vascular aging in humans. Hypertension. 2010 Feb;55(2):319-26. doi: 10.1161/HYPERTENSIONAHA.109.141275. Epub 2010 Jan 11. PMID 20065154
- [Background] Redheuil A, Yu WC, Mousseaux E, Harouni AA, Kachenoura N, Wu CO, Bluemke D, Lima JA. Age-related changes in aortic arch geometry: relationship with proximal aortic function and left ventricular mass and remodeling. J Am Coll Cardiol. 2011 Sep 13;58(12):1262-70. doi: 10.1016/j.jacc.2011.06.012. PMID 21903061
- [Background] Rosenbaum D, Koch E, Girerd X, Rossant F, Paques M. [Imaging of retinal arteries with adaptative optics, feasibility and reproducibility]. Ann Cardiol Angeiol (Paris). 2013 Jun;62(3):184-8. doi: 10.1016/j.ancard.2013.04.017. Epub 2013 May 29. French. PMID 23773704
- [Background] Herment A, Kachenoura N, Lefort M, Bensalah M, Dogui A, Frouin F, Mousseaux E, De Cesare A. Automated segmentation of the aorta from phase contrast MR images: validation against expert tracing in healthy volunteers and in patients with a dilated aorta. J Magn Reson Imaging. 2010 Apr;31(4):881-8. doi: 10.1002/jmri.22124. PMID 20373432
- [Background] Bollache E, Kachenoura N, Redheuil A, Frouin F, Mousseaux E, Recho P, Lucor D. Descending aorta subject-specific one-dimensional model validated against in vivo data. J Biomech. 2014 Jan 22;47(2):424-31. doi: 10.1016/j.jbiomech.2013.11.009. Epub 2013 Nov 15. PMID 24290136
- [Background] Dogui A, Kachenoura N, Frouin F, Lefort M, De Cesare A, Mousseaux E, Herment A. Consistency of aortic distensibility and pulse wave velocity estimates with respect to the Bramwell-Hill theoretical model: a cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2011 Jan 27;13(1):11. doi: 10.1186/1532-429X-13-11. PMID 21272312